CLINICAL TRIAL: NCT04452864
Title: Can a Serious Game-based Cognitive Training Attenuate Cognitive Decline Related to Alzheimer's Disease
Brief Title: Tablet-based Cognitive Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2020-00630
Record Dates: First submitted 2020-06-24; First posted 2020-07-01 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Alzheimer Disease; Dementia; Mild Cognitive Impairment
Keywords: Alzheimer Disease; Dementia; Mild Cognitive Impairment; Cognitive Training; Serious Games
MeSH Terms: conditions — Alzheimer Disease; Dementia; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of three study arms and conduct a Computerized Cognitive Training (CCT) at home (daily) and on site (weekly) for 10 weeks. Before and after the CCT, neuropsychological assessments will be conducted.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Study Intervention (Experimental): The study intervention consists of a tablet-based cognitive training, targeting the cognitive domains mostly affected by AD. This training will be performed for three months (each day for 20 minutes). After three months this group will continue the training at home for six months and meet monthly for group sessions (i.e. booster sessions) on site.
  Interventions: Device: Computerized Cognitive Training
- Active Control Group (Active Comparator): This control study arm will watch documentaries at home for three months (each day for 20 minutes) , instead of performing the CCT and serve as active control group. This group will also train with the CCT tasks after these three months.
  Interventions: Device: Documentaries with delayed Computerized Cognitive Training
- Wait-List Control (Other): This control study arm will start with the CCT with a delay of three months and serve as wait-list control group.
  Interventions: Device: Computerized Cognitive Training

INTERVENTIONS:
Device: Computerized Cognitive Training — The study intervention consists of a tablet-based cognitive training, targeting the cognitive domains mostly affected by Alzheimer Disease.
  Arms: Study Intervention; Wait-List Control
Device: Documentaries with delayed Computerized Cognitive Training — The active control group watches documentaries for three months before starting with the CCT.
  Arms: Active Control Group

SUMMARY:
Today the therapy options for dementia due to Alzheimer's disease (AD) are limited. One recommended intervention is cognitive stimulation. We try to develop serious games as a further treatment option, also usable in pre-dementia as well as early stages of dementia and for a long period of time.

The main objective of this study is to test, if the computerized-cognitive training (CCT) is able to improve the performance in a score quantifying an "AD-specific" component score. Additionally, the neurobiological effects of the training are investigated.

DETAILED DESCRIPTION:
The study intervention consists of a computer-based cognitive training, targeting the cognitive domains mostly affected by AD. This training will be performed for three months (each day for 20 minutes). After three months the intervention group will continue the training at home for six months and meet monthly for group sessions (i.e. booster sessions) on site.

Primary endpoint will be the change in an "AD-specific" component score, quantified by episodic memory, semantic memory and visuospatial abilities. Secondary endpoints are changes in task related brain networks and changes in resting state networks.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Alzheimer's Disease
* Patients with increased risk for developing dementia
* Must be able to give their consent

Exclusion Criteria:

* Contra-indications for MRI scanning
* Substance abuse
* Severe medical conditions

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2024-07-09 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Change in AD specific component score | The primary endpoint will be assessed four times, with breaks of three months in between. Primary outcome will be assessed up to 9 months.
  The outcome is quantified by an AD component score including measures of EM (auditory verbal learning), SM (verbal fluency, naming task) and spatial abilities (Rey-Osterrieth complex figure test). These scores will be assessed four times, before the training as well as after three, six and nine months by tablet-based cognitive tests. A short follow-up assessment will be performed after a total of 12 months which does not include primary outcome measure.

SECONDARY OUTCOMES:
MRI functional and structural | Secondary endpoints will be assessed two to four times, depending on the study arm, as MRI assessments are not always performed after six and nine months.
  Secondary endpoints are changes in task related brain networks (i.e. spatial ability and episodic memory) and changes in resting state networks.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Klöppel, Prof. Dr., Principal Investigator — University of Bern
Locations (2):
- Switzerland (2):
  - University Hospital of Old Age Psychiatry and Psychotherapy, Bern
  - Memory Clinic Zentralschweiz, Lucerne

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication will be published pseudonymized in a open access data base
Time Frame: IPD and any additional material will be available when data collection and analysis is completed Items will be retained for the lifetime of the repository (at least 20years)
Access Criteria: According to SNF Guidelines IPD will be published in a open access data base

REFERENCES:
- [Background] Brill E, Krebs C, Falkner M, Peter J, Henke K, Zust M, Minkova L, Brem AK, Kloppel S. Can a serious game-based cognitive training attenuate cognitive decline related to Alzheimer's disease? Protocol for a randomized controlled trial. BMC Psychiatry. 2022 Aug 12;22(1):552. doi: 10.1186/s12888-022-04131-7. PMID 35962371